CLINICAL TRIAL: NCT01246466
Title: Feasibility Trial of a Hybrid Approach for Treatment of Patients With Persistent or Longstanding Persistent Atrial Fibrillation With Radiofrequency Ablation
Brief Title: Dual Epicardial Endocardial Persistent Atrial Fibrillation (AF) Study
Acronym: DEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP2009-1
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Results first posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2016-01

CONDITIONS: Persistent Atrial Fibrillation; Longstanding Persistent Atrial Fibrillation
Keywords: Persistent Atrial Fibrillation; Longstanding Persistent Atrial Fibrillation; Ablation; Catheter ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AtriCure Bipolar System combined with a catheter ablation (Experimental): procedure using the AtriCure Bipolar System plus a catheter ablation
  Interventions: Device: Hybrid: AtriCure Bipolar System & EP ablation procedure

INTERVENTIONS:
Device: Hybrid: AtriCure Bipolar System & EP ablation procedure — AtriCure Bipolar System plus a catheter ablation

SUMMARY:
The purpose of this clinical investigation is to evaluate how safe a less invasive cardiac surgery is using the AtriCure Bipolar System combined with a catheter ablation procedure in treating AF, and how effective this combined procedure is using the AtriCure System in treating AF. The AtriCure Bipolar System will be used to perform the less invasive cardiac surgery and a standard electrophysiology catheter, currently available, will be used to perform the catheter ablation procedure. This surgical procedure is considered less invasive because it is done through tiny surgical punctures on the sides of the chest near the ribs instead of one large surgical incision of the breast bone to completely open the chest and access the heart, and it also avoids the need for the heart-lung bypass machine.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Patients with symptomatic (e.g. palpitations, shortness of breath, fatigue) persistent or longstanding persistent AF Persistent
3. Patient is willing and able to provide written informed consent.
4. Patient has a life expectancy of at least 2 years.
5. Patient is willing and able to attend the scheduled follow-up visits.

Exclusion Criteria:

1. Prior Cardiothoracic Surgery.
2. Patient has NYHA Class IV heart failure.
3. Evidence of underlying structural heart disease requiring surgical treatment.
4. Ejection fraction < 30%
5. Measured left atrial diameter > 6.0 cm
6. Renal Failure
7. Stroke within previous 6 months.
8. Known carotid artery stenosis greater than 80%.
9. Evidence of significant active infection or endocarditis.
10. Pregnant woman or women desiring to become pregnant in the next 24 months.
11. Presence of thrombus in the left atrium determined by echocardiography.
12. History of blood dyscrasia.
13. Contraindication to anticoagulation, based on Investigator's opinion.
14. Mural thrombus or tumor.
15. Moderate to Severe COPD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Stanford University Medical Center, Stanford, California
  - Vanderbilt Heart Institute, Nashville, Tennessee
  - Baylor Health, Plano, Texas
  - UVA, Charlottesville, Virginia
  - Sentara Norfolk, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 5 academic medical centers. The first participant was enrolled in December 2010 and the last participant was enrolled in October 2011.
Groups:
- AtriCure Bipolar System Combined With a Catheter Ablation: Procedure using the AtriCure Bipolar System plus a catheter ablation
  Hybrid ablation procedure: AtriCure Bipolar System plus a catheter ablation
Period: Overall Study
Arm/Group | AtriCure Bipolar System Combined With a Catheter Ablation
Started | 24
Completed | 22
Not Completed | 2
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | AtriCure Bipolar System Combined With a Catheter Ablation
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24
Height [Mean (Standard Deviation); unit: inches] | 70.5 (2.9)
Weight [Mean (Standard Deviation); unit: pounds] | 214.7 (33.4)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.4 (4.2)

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint
Description: Acute MAE within 30 days post procedure or hospital discharge (up to 7 days), whichever is longer.
Time Frame: Within the first 30 days post-index procedure, or hospital discharge (up to 7 days), whichever is longer.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AtriCure Bipolar System Combined With a Catheter Ablation
Number analyzed (Participants) | 24
percentage of participants
  Death per IPA | 0 [0.0 to 14.2]
  Excessive bleeding per IPA | 0 [0.0 to 14.2]
  Stroke per IPA | 4.2 [0.1 to 21.1]
  TIA per IPA | 0 [0.0 to 14.2]
  MI per IPA | 4.2 [0.1 to 21.1]
  Cardiac Tamponade per IPA | 0 [0.0 to 14.2]
  Pulmonary Embolism per IPA | 0 [0.0 to 14.2]
  Peripheral Embolism per IPA | 0 [0.0 to 14.2]
  Atrio-esophageal Fistula per IPA | 0 [0.0 to 14.2]
  Diaphragmatic Paralysis per IPA | 0 [0.0 to 14.2]
  Pulmonary Vein Stenosis per IPA | 0 [0.0 to 14.2]
  New 2nd/3rd Degree AV Block Requiring PPM per IPA | 0 [0.0 to 14.2]
  Serious Skin Burns per IPA | 0 [0.0 to 14.2]
  Conversion to Thoracotomy or Sternotomy per IPA | 8.3 [1.0 to 27.0]
  Catheter Related SAEs per IPA | 12.5 [2.7 to 32.4]
  Surgical Procedure Related SAEs per IPA | 20.8 [7.1 to 42.2]
  Death per FDA | 0 [0.0 to 14.2]
  Excessive Bleeding per FDA | 0 [0.0 to 14.2]
  Stroke per FDA | 4.2 [0.1 to 21.1]
  TIA per FDA | 0 [0.0 to 14.2]
  MI per FDA | 4.2 [0.1 to 21.1]
  Cardiac Tamponade per FDA | 0 [0.0 to 14.2]
  Pulmonary Embolism per FDA | 0 [0.0 to 14.2]
  Atrioesophageal Fistula per FDA | 0 [0.0 to 14.2]
  Diaphragmatic Paralysis per FDA | 0 [0.0 to 14.2]
  Pulmonary Vein Stenosis per FDA | 0 [0.0 to 14.2]
  New 2nd/3rd Degree AV Block Requiring PPM per FDA | 0 [0.0 to 14.2]
  Serious Skin Burns per FDA | 0 [0.0 to 14.2]
  Conversion to Thoracotomy or Sternotomy per FDA | 8.3 [1.0 to 27.0]
  Catheter Related SAEs per FDA | 8.3 [1.0 to 27.0]

2. Primary Outcome: Absence of Atrial Fibrillation
Description: Absence of atrial fibrillation (AF) at twelve month follow-up based on an auto trigger event monitor, while off all Class I and III antiarrhythmic therapy.
Time Frame: 12 month follow-up
Population: Denominators (19) are subjects who are evaluable for primary efficacy endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AtriCure Bipolar System Combined With a Catheter Ablation
Number analyzed (Participants) | 19
percentage of participants
  Success at 12 Months | 68.4 [43.4 to 87.4]
  Failure by AAD | 10.5 [1.3 to 33.1]
  Failure by Holter/Pacemaker Interrogation | 21.1 [6.1 to 45.6]
  Atrial Fibrillation | 0.0 [0.0 to 17.6]
  Atrial Flutter | 0 [0.0 to 17.6]
  Atrial Tachycardia | 21.1 [6.1 to 45.6]
  Failure by both AAD and Holter/Pacemaker Interrog | 0.0 [0.0 to 17.6]

3. Secondary Outcome: Overall Serious Device or Procedure Related Adverse Event Rate
Time Frame: 12 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | AtriCure Bipolar System Combined With a Catheter Ablation
Number analyzed (Participants) | 24
Participants
  Excessive Bleeding | 0
  Stroke | 1
  TIA | 0
  MI | 1
  Cardiac Tamponade | 0
  Pulmonary Embolism | 0
  Peripheral Embolism | 0
  Atrio-esophageal Fistula | 0
  Diaphragmatic Paralysis | 0
  Pulmonary Vein Stenosis | 0
  New 2nd/3rd Degree AV Block Requiring PPM | 0
  Serious Skin Burns | 0
  Conversion to Thoracotomy or Sternotomy | 2
  Catheter Related SAEs | 2
  Surgical Procedure Related SAEs | 0

4. Secondary Outcome: Acute Procedure Success
Time Frame: Upon completion of the index procedure, up to ten hours
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AtriCure Bipolar System Combined With a Catheter Ablation
Number analyzed (Participants) | 24
percentage of participants
  Inferior Right Pulmonary Veins Isolation Evaluated | 100 [85.8 to 100.0]
  Inferior Right Pulmonary Veins Isolation Achieved | 100 [85.8 to 100.0]
  Inferior Left Pulmonary Veins Isolation Evaluated | 100 [85.8 to 100.0]
  Inferior Left Pulmonary Veins Isolation Achieved | 95.8 [78.9 to 99.9]
  Superior Right Pulmonary Veins Isolation Evaluated | 100.0 [85.8 to 100.0]
  Superior Right Pulmonary Veins Isolation Achieved | 100.0 [85.8 to 100.0]
  Superior Left Pulmonary Veins Isolation Evaluated | 100.0 [85.8 to 100.0]
  Superior Left Pulmonary Veins Isolation Achieved | 100.0 [85.8 to 100.0]
  Left Atrium Posterior Box Isolation Evaluated | 100.0 [85.8 to 100.0]
  Left Atrium Posterior Box Isolation Achieved | 54.2 [32.8 to 74.4]
  Bi-drectional block Mitral Valve Isthmus Evaluated | 100.0 [85.8 to 100.0]
  Bi-drectional block Mitral Valve Isthmus Achieved | 83.3 [62.6 to 95.3]
  Bi-directional block of RC isthmus evaluated | 100.0 [85.8 to 100.0]
  Bi-directional block of RC isthmus achieved | 83.3 [62.6 to 95.3]
  Superior Vena Cava block evaluated | 100.0 [85.8 to 100.0]
  Superior Vena Cava block achieved | 87.5 [67.6 to 97.3]

5. Secondary Outcome: Absence of Atrial Fibrillation
Description: Absence of atrial fibrillation after the 3 month blanking period through twelve month follow-up based on auto trigger event monitor.
Time Frame: After the 3 month blanking period through twelve month follow-up.
Population: Denominators are subjects who are evaluable for secondary efficacy endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | AtriCure Bipolar System Combined With a Catheter Ablation
Number analyzed (Participants) | 24
Participants
  Efficacy Evaluable at 6 months | 22
  Free of AF independent of the need for AADs at 6M: number analyzed (Participants) | 22
  Free of AF independent of the need for AADs at 6M | 20
  Efficacy Evaluable at 12 Months | 19
  Free of AF independent of the need for AADs at 12M: number analyzed (Participants) | 19
  Free of AF independent of the need for AADs at 12M | 15

6. Secondary Outcome: Number of Participants With Reintervention to Address Atrial Dysrhythmia
Description: Number of Participants with Reintervention to Address Atrial Dysrhythmia, through 12 months
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | AtriCure Bipolar System Combined With a Catheter Ablation
Number analyzed (Participants) | 24
Participants | 2

7. Secondary Outcome: Number of Participants With DC Cardioversion
Time Frame: 12 months
Reporting Status: Not Posted

8. Secondary Outcome: Improvement in AF
Description: Improvement in Atrial Fibrillation Symptom Checklist Frequency (Minimum value: -1.0, Maximum value: 25.0) and Severity Scores (Minimum value: -6.0, Maximum value: 19.0)
Time Frame: 12 months
Population: Denominators are subjects who are evaluable for secondary efficacy endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AtriCure Bipolar System Combined With a Catheter Ablation
Number analyzed (Participants) | 24
units on a scale
  Change in AF Symptom Checklist Frequency Score: number analyzed (Participants) | 22
  Change in AF Symptom Checklist Frequency Score | 13.4 (8.4)
  Change in AF Symptom Checklist Severity Score: number analyzed (Participants) | 21
  Change in AF Symptom Checklist Severity Score | 9.8 (7.2)

9. Secondary Outcome: Duration of Procedure
Time Frame: During index procedure
Population: Denominators are subjects who are evaluable for secondary efficacy endpoint.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | AtriCure Bipolar System Combined With a Catheter Ablation
Number analyzed (Participants) | 24
Hours
  Total Surgery Time | 8.9 (1.2)
  Epicardial Surgical Procedure Time | 3.9 (0.9)
  EP Catheter Procedure Time: number analyzed (Participants) | 23
  EP Catheter Procedure Time | 2.9 (1.1)

ADVERSE EVENTS:
Time Frame: Treatment to 24 months
Arm/Group | AtriCure Bipolar System Combined With a Catheter Ablation
Serious Adverse Events (participants affected / at risk) | 16/24
Other Adverse Events (participants affected / at risk) | 20/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AtriCure Bipolar System Combined With a Catheter Ablation (N=24)
Embolic Stroke (Nervous system disorders) | 1 (1)
Cardiac Perforation (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1)
Embolic Stroke - Epicardial Ablation Procedure (Nervous system disorders) | 1 (1)
Vocal Cord Paresis (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Neuropathy Peripheral (Nervous system disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Mediastinal Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial Fibrillation - Other Relationship (Cardiac disorders) | 2 (2)
Atrial Flutter - Other Relationship (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 3 (3)
Ventricular Fibrillation - Other Relationship (Cardiac disorders) | 1 (2)
Visual Impairment (Eye disorders) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Implantable Defribrillator Malfunction (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Ischaemia (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AtriCure Bipolar System Combined With a Catheter Ablation (N=24)
Embolic Stroke (Nervous system disorders) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1)
Cardiac Perforation (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1)
Cardiac Vein Perforation (Injury, poisoning and procedural complications) | 1 (1)
Embolic Stroke - Epicardial Ablation Procedure (Nervous system disorders) | 1 (1)
Vocal Cord Paresis (Nervous system disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Pericarditis (Cardiac disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Mouth Ulceration (Gastrointestinal disorders) | 1 (1)
Postoperative Ileus (Injury, poisoning and procedural complications) | 1 (1)
Neuropathy Peripheral (Nervous system disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Mediastinal Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anaemia - Other Relationship (Blood and lymphatic system disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 2 (2)
Atrial Flutter - Other Relationship (Cardiac disorders) | 1 (1)
Atrioventricular Block (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 3 (4)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Ventricular Fibrillation (Cardiac disorders) | 1 (2)
Hypothyroidism (Endocrine disorders) | 1 (1)
Visual Impairment (Eye disorders) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 1 (1)
Chest Pains (General disorders) | 2 (3)
Non-Cardiac Chest Pain (General disorders) | 1 (2)
Oedema Peripheral (General disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 4 (4)
Implantable Defribillator Malfunction (Injury, poisoning and procedural complications) | 1 (1)
Ulnar Nerve Injury (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1)
Essential Tremor (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 1 (1)
Ischaemia (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes